CLINICAL TRIAL: NCT00398151
Title: An Open-Label Study to Evaluate the Inflammatory Markers in Adult Patients With Asthma Associated With Allergic Rhinitis Receiving Montelukast Therapy
Brief Title: To Evaluate the Inflammatory Markers in Adult Patients With Asthma Associated With Allergic Rhinitis Receiving Montelukast Therapy (0476-366)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0476-366; 2006_043
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Duration of Therapy

INTERVENTIONS:
Drug: MK0476, montelukast sodium / Duration of Treatment: 12 Weeks

SUMMARY:
To evaluate the changes in proinflammatory markers (ltd4 in urine) and eosinophil from peripheral blood after newly initiated montelukast therapy.

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis symptoms: sneezing, rhinorrhea, obstruction of the nasal passages, itchy nose and throat, and conjunctival
* Male or female outpatient 20 years of age and older
* Patients with the following signs and symptoms of asthma and allergic rhinitis: history of cough, wheezing, shortness of breath, positive methacholine bronchoprovocation test

Exclusion Criteria:

* Active, acute or chronic, pulmonary disorder (besides asthma) documented by history, physical examination, or chest x-ray. history of anaphylactic or hypersensitive to study drug
* Requires oral, intravenous, or intramuscular corticosteroids on daily routine basis
* Started on immunotherapy within six months before the pre-study visit and/or the dose of immunotherapy is expected to change over the course of the study
* Treated with montelukast within 3 months before enrollment
* Unable to perform acceptable, reproducible spirometry and peak flow measurement
* Unresolved symptoms and signs of an upper respiratory tract infection (uri) within 2 weeks prior to visit 1

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-08-01 (Actual); Primary Completion 2006-01-18 (Actual); Study Completion 2006-01-18 (Actual)

PRIMARY OUTCOMES:
Ltd4 in urine and eosinophil from peripheral blood over 3 months of therapy

SECONDARY OUTCOMES:
Asthma symptoms score throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC